CLINICAL TRIAL: NCT04333082
Title: Refractory Status Epilepticus Treatment (RESET): Quality and Efficacy of Coma Induction
Brief Title: Refractory Status Epilepticus Treatment: Quality and Efficacy of Coma Induction
Acronym: RESET
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00538; me20Sutter
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Status Epilepticus; Refractory Status Epilepticus
Keywords: artificial deep coma; intravenous anesthetic drugs (IVADs); total seizure oppression
MeSH Terms: conditions — Status Epilepticus | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — collection of patient data
  Data collection (demographics, prehospital management, duration of ICU and hospital stay, destination at discharge, date(s) of seizure(s), electroencephalographic (EEG) data, seizure history and etiology, number and duration of SE episodes, medication, types of SE according to the current guidelines from the International League of Epilepsy (ILAE), neuroimaging features, comorbidities, laboratory parameters, complications during and after SE , laboratory testing, vital signs, fluid balance) will be performed from the digital medical records, the electroencephalographic and microbiologic database of patients

SUMMARY:
This study is to investigate the effects of different treatment characteristics regarding the use of intravenous anesthetic drugs (IVADs) as a rescue treatment for refractory Status epilepticus (RSE) on course and outcome. A retrospective data extraction from the digital medical records, the electroencephalographic and microbiologic database of all consecutive adult patients with Status epilepticus (SE) admitted to the University Hospital Basel is undertaken.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed SE between 2005 and 2019 who have been treated at intensive care units (ICUs) of the University Hospital of Basel

Exclusion Criteria:

* Patients with repetitive epileptic seizures not qualifying for SE or RSE
* Patients with documented refusal of the general in-house consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (i.e., patients ≥18 years of age) with diagnosed SE between 2005 and 2019 who have been treated at intensive care units (ICUs) of the University Hospital of Basel, a Swiss tertiary academic medical care center
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
number of in- hospital death | at baseline (T0)
  number of in- hospital death

SECONDARY OUTCOMES:
neurofunctional alteration assessed by Glasgow Outcome Score (GOS) | at baseline (T0)
  neurofunctional alteration assessed by Glasgow Outcome Score (GOS). The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories: Dead, Vegetative State, Severe Disability, Moderate Disability or Good Recovery

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, PD Dr. med, Principal Investigator — Universitätsspital Basel / Intensivmedizin
Locations (1):
- Clinic for Intensive Care Medicine, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Fisch U, Junger AL, Baumann SM, Semmlack S, De Marchis GM, Hunziker S, Ruegg S, Marsch S, Sutter R. Association Between Induced Burst Suppression and Clinical Outcomes in Patients With Refractory Status Epilepticus: A 9-Year Cohort Study. Neurology. 2023 May 9;100(19):e1955-e1966. doi: 10.1212/WNL.0000000000207129. Epub 2023 Mar 8. PMID 36889924